CLINICAL TRIAL: NCT04784416
Title: Transcranial Photobiomodulation for Alzheimer's Disease (TRAP-AD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Alzheimer's Association (Other); LiteCure LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-00865
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Transcranial Photobiomodulation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcranial Photobiomodulation (t-PBM) (Experimental)
  Interventions: Device: Active tPBM-2.0; Drug: 18F-MK-6240
- Sham (Sham Comparator)
  Interventions: Device: Sham tPBM-2.0; Drug: 18F-MK-6240

INTERVENTIONS:
Device: Active tPBM-2.0 — The NIR continuous wave (average irradiance = 300 mW/cm2) will be used. The duration or irradiation will be for ~11 minutes (666 seconds).
  Arms: Transcranial Photobiomodulation (t-PBM)
Device: Sham tPBM-2.0 — The sham mode (0 mW/cm2) will be used. The duration or sham "irradiation" will be for ~11 minutes (666 seconds).
  Arms: Sham
Drug: 18F-MK-6240 — PET tracer to be injected prior to PET imaging session, which will occur during baseline assessments

SUMMARY:
This multi-site study will be the first to evaluate the dose-dependent effects of t-PBM in amnestic Mild Cognitive Impairment (aMCI) and early Alzheimer's Disease (AD) (CDR of 0.5-1, FAST 1-4; age 65-85) in a randomized clinical trial of 8 weeks of t-PBM vs. sham. At baseline, all subjects will complete initial neuropsychological testing. To elucidate mechanisms of action of t-PBM, prior to treatment, subjects will undergo neuroimaging related to critical features of AD: tau 18F MK-6240 load (PET), measures of brain bioenergetics (31P-MRS), and functional connectivity (rs-fMRI). After undergoing target engagement testing (t-PBM session performed during fMRI to detect BOLD changes with active t-PBM), subjects will then be randomized to t-PBM/sham and complete 24 t-PBM/sham treatments, ~11 min per day, 3 days per week, for 8 weeks. t-PBM will be administered via continuous, 808 nm wavelength laser delivery to the forehead bilaterally (at standard EEG electrode positions F4, F3).

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and follow study procedures.
2. Age > or = 65 years and < or = 85 years.
3. Meets the Petersen MCI criteria for Amnestic MCI (single and multiple domain) with a Clinical Dementia Rating (CDR) between 0.5-1.0, and a Functional Assessment Staging (FAST) of 1-4.
4. Be willing to identify an informed relative, family member, spouse, or friend for study staff to interview to confirm subject reports as per UDS 3.0 guidelines; however the lack of a study informant is not exclusionary.
5. Have at least a high school diploma/12 years of education.
6. Participants with current mild MDD may be allowed to participate, given that mild MDD does not affect cognition and does not pose increased risk to the participant, as determined by site PI on a case-by-case basis.

Exclusion Criteria:

1. Unwilling/unable to comply with study procedures.
2. Other diagnosis of dementia (i.e. not Alzheimer's type), history of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, intellectual disability, or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders).
3. History of significant cerebrovascular pathology (e.g., significant stroke). Subjects with a history of cardiovascular disease (e.g., myocardial infarction) will be allowed to participate at site PI's discretion, on a case-by-case basis, given that the cardiovascular disease is stable and does not reflect the presence of significant cerebrovascular pathology.
4. Clinically unstable systemic medical disorders.
5. Current DSM-5 diagnosis of alcohol or drug use disorder or other major psychiatric illness (e.g., schizophrenia, bipolar, PTSD, depression). Participants with current mild MDD may be allowed to participate, given that mild MDD does not affect cognition and does not pose increased risk to the participant, as determined by site PI on a case-by-case basis. Participants with current moderate/severe MDD will be excluded.
6. Clinical or laboratory evidence of hypothyroidism.
7. Clinically significant abnormal findings of laboratory parameters or at physical examination.
8. Medications affecting cognition (e.g., narcotic analgesics; chronic use of medications with anticholinergic activity, anti-Parkinsonian medications, antipsychotic meds, etc.). Stable use (i.e., = 6 months) of memantine or acetylcholinesterase inhibitors will be allowed.
9. Family history of early onset (<60 y/o) dementia.
10. Past intolerance or hypersensitivity to t-PBM.
11. Significant skin conditions on the subject's scalp in the area of the procedure sites.
12. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.
13. Any type of implants in the head, whose functioning might be affected by t-PBM.
14. The completion of study imaging procedures is highly encouraged, but not mandatory for participants with extenuating circumstances (e.g., having prosthetic devices or metallic foreign bodies that constitute hazards for MRI, unable to get PET due to previous level of radiation exposure, having claustrophobia, having a large body size and shape).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) Total Scale Index Score. | Baseline, Week 8
  RBANS is s a brief, individually administered battery to measure cognitive decline or improvement. Total Scale Index Score Range = 40-160. A higher score indicates better performance.

SECONDARY OUTCOMES:
Change in Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) Total Scale Index Score. | Baseline, Month 3
  RBANS is s a brief, individually administered battery to measure cognitive decline or improvement. Total Scale Index Score Range = 40-160. A higher score indicates better performance.
Addenbrooke's Cognitive Examination (ACE-III) Score | Baseline
  ACE-III is a screening test that is composed of tests of attention, orientation, memory, language, visual perceptual and visuospatial skills. The total range of raw score is 0-100. A higher score indicates more intact cognitive functioning.
Addenbrooke's Cognitive Examination (ACE-III) Score | Week 8
  ACE-III is a screening test that is composed of tests of attention, orientation, memory, language, visual perceptual and visuospatial skills. The total range of raw score is 0-100. A higher score indicates more intact cognitive functioning.
Addenbrooke's Cognitive Examination (ACE-III) Score | Month 3
  ACE-III is a screening test that is composed of tests of attention, orientation, memory, language, visual perceptual and visuospatial skills. The total range of raw score is 0-100. A higher score indicates more intact cognitive functioning.
Letter Comparison Test Score | Baseline
  The total range of score is 0-21. A higher raw score indicates better performance.
Letter Comparison Test Score | Week 8
  The total range of score is 0-21. A higher raw score indicates better performance.
Letter Comparison Test Score | Month 3
  The total range of score is 0-21. A higher raw score indicates better performance.
Pattern Comparison Test Score | Baseline
  The total range of score is 0-30. A higher raw score indicates better performance.
Pattern Comparison Test Score | Week 8
  The total range of score is 0-30. A higher raw score indicates better performance.
Pattern Comparison Test Score | Month 3
  The total range of score is 0-30. A higher raw score indicates better performance.
Stroop Color and Word Test (SCWT) | Baseline
  SCWT is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. This study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Stroop Color and Word Test (SCWT) | Week 8
  SCWT is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. This study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Stroop Color and Word Test (SCWT) | Month 3
  SCWT is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. This study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Difference in Score Between Trail Making Test-A (TMT-A) and Trail Making Test-B (TMT-B) | Baseline
  Trails Making Test (Trails) is a neuropsychological test of visual attention and task switching. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1-25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); as in Part A, the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time it takes to connect the "trail" is recorded.
  Reported as B - A. Range = 0 - 100+ (measured in seconds). A higher B - A score indicates poorer performance.
Difference in Score Between Trail Making Test-A (TMT-A) and Trail Making Test-B (TMT-B) | Week 8
  Trails Making Test (Trails) is a neuropsychological test of visual attention and task switching. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1-25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); as in Part A, the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time it takes to connect the "trail" is recorded.
  Reported as B - A. Range = 0 - 100+ (measured in seconds). A higher B - A score indicates poorer performance.
Difference in Score Between Trail Making Test-A (TMT-A) and Trail Making Test-B (TMT-B) | Month 3
  TMT is a neuropsychological test of visual attention and task switching. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1-25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); as in Part A, the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time it takes to connect the "trail" is recorded.
  Reported as B - A. Range = 0 - 100+ (measured in seconds). A higher B - A score indicates poorer performance.
TMT-B T-Score | Baseline
  In TMT-B, the circles include both numbers (1-13) and letters (A-L); the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time is takes to connect the "trail" is recorded. Range = 0 - 100. A higher T-score indicates better performance
TMT-B T-Score | Week 8
  In TMT-B, the circles include both numbers (1-13) and letters (A-L); the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time is takes to connect the "trail" is recorded. Range = 0 - 100. A higher T-score indicates better performance
TMT-B T-Score | Month 3
  In TMT-B, the circles include both numbers (1-13) and letters (A-L); the patient draws lines to connect the circles in an ascending pattern (alternating numbers and letters). The time is takes to connect the "trail" is recorded. Range = 0 - 100. A higher T-score indicates better performance
Face-Name Associative Memory Exam (FNAME-12) Score | Baseline
  FNAME-12 is an associative memory test where participants see a series of facial photos and names and are asked to remember the face-name pairs.
Face-Name Associative Memory Exam (FNAME-12) Score | Week 8
  FNAME-12 is an associative memory test where participants see a series of facial photos and names and are asked to remember the face-name pairs.
Face-Name Associative Memory Exam (FNAME-12) Score | Month 3
  FNAME-12 is an associative memory test where participants see a series of facial photos and names and are asked to remember the face-name pairs.
Letter Number Sequencing Score | Baseline
  this study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Letter Number Sequencing Score | Week 8
  this study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Letter Number Sequencing Score | Month 3
  this study will use T-scores, range = 20 - 80. A higher T-score indicates better performance.
Change in Systemic Assessment for Treatment Emergent Events - Specific Inquiry (SAFTEE-SI) Score | Baseline, up to Week 8
  SAFTEE-SI is a list of 55 symptoms. Participants indicate how bothersome each symptom has been for them by circling the appropriate number (0-none, 1-mild, 2-moderate, 3-severe). The total range of score is 0 - 165. The higher the score, the more severely bothersome the symptoms are.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, Principal Investigator — NYU Langone Health and Nathan Kline Institute; Ricardo Osorio, MD, Principal Investigator — NYU Langone Health and Nathan Kline Institute; Paolo Cassano, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be provided upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access upon reasonable request.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04784416/ICF_000.pdf